CLINICAL TRIAL: NCT05774665
Title: Specialized Pro-resolving Lipid Mediators and Treatment Resistant Depression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Utah (Other); Emory University (Other)
Responsible Party: Principal Investigator, David Mischoulon, MD, PhD, Director, Depression Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R33AT012329 (NIH)
Record Dates: First submitted 2023-03-06; First posted 2023-03-20 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Treatment Resistant Depression; Inflammation; Overweight
Keywords: omega-3; fatty acid; major depressive disorder
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Inflammation; Overweight; Depressive Disorder, Major | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Intervention Model Description: Double blind randomized placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study will be placebo controlled. Participants will receive identical capsules with omega-3 fatty acids or placebo. Randomization will be set by our research pharmacy and no participants or study personnel will know treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Omega-3 (Experimental): Omega-3 fatty acid (ProEPA Xtra) capsules containing a total of 4 g/day of eicosapentaenoic acid (EPA), administered for 12 weeks.
  Interventions: Drug: Omega 3
- Placebo (Placebo Comparator): Placebo capsules containing soybean oil (about 54% omega-6 and 6% omega-3, but no EPA or docosahexaenoic acid (DHA)), and matched to the ProEPA Xtra capsules in terms of appearance, odor, and taste.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Omega 3 — Omega-3 fatty acid enriched for eicosapentaenoic acid (EPA)
  Other Names: EPA
  Arms: Omega-3
Other: Placebo — Placebo consisting of soybean oil (about 54% omega-6 and 6% omega-3, but no EPA or docosahexaenoic acid (DHA)).
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to determine the impact of omega-3 fatty acids on the production of anti-inflammatory effects and clinical improvement in people with depression who have not responded well to standard antidepressant treatment. The main questions it seeks to answer are:

1. Do omega-3 fatty acids added to ineffective antidepressant treatment increase production of compounds that reduce inflammation?
2. Is the increase in these anti-inflammatory compounds associated with a stronger antidepressant effect?

Participants taking antidepressants that have not worked completely will be assigned at random for a 12-week period to one of the following:

1. an omega-3 preparation
2. an inactive placebo

During the course of the study, blood tests will be obtained for compounds associated with inflammation, and questionnaires to measure clinical improvement in depressive symptoms will be administered.

DETAILED DESCRIPTION:
This R33 application builds directly on a previous collaborative R01 (NCT00517036) and UG3 (NCT02553915) grants. The investigators will carry out a 12-week, randomized placebo-controlled, double-masked, augmentation trial of 4 g/day eicosapentaenoic acid (EPA)-enriched omega-3 treatment in adults with major depressive disorder (MDD), an inadequate response to antidepressants (treatment-resistant depression [TRD]), body mass index (BMI) >25 kg/m2 and ≤ 40 kg/m2, and inflammation (high sensitivity C reactive protein [hs-CRP] ≥ 3 mg/L and ≤ 10 mg/L). It is hypothesized that 4 g/day of EPA-enriched omega-3 will: 1) Significantly increase plasma 18-hydroxy eicosapentaeoic acid [18-HEPE] concentrations compared to placebo (primary biological endpoint); 2) produce significantly greater increases in plasma 18-HEPE concentration since baseline for sustained MADRS responders (those with at least 50% reduction since baseline in MADRS scores at both treatment week 8 and week 12) than for (a) unsustained/non-responders to EPA-enriched n-3 as well as (b) placebo-supplemented sustained responders (secondary biological endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years
* Patients with treatment-resistant MDD who have not responded to at least 2 and no more than 5 antidepressant trials of at least 8 weeks duration during the current episode and have been on a current stable antidepressant regiment for at least 4 weeks. The diagnosis of MDD will be confirmed using the MINI and the historical failure to respond to antidepressant therapy will be documented using the Antidepressant Treatment Response Questionnaire (ATRQ), with failure to respond defined as less than 50% improvement by subject history.
* hs-CRP ≥ 3 mg/L and ≤ 10 mg/L
* BMI >25 kg/m2 and ≤ 40 kg/m2
* 17-item Hamilton Depression Rating Scale (HAM-D) score ≥15, and <25% decrease in score between screen and baseline

Exclusion Criteria:

Diagnostic Exclusions:

* Meeting lifetime DSM-5 criteria for: a neurocognitive disorder, psychotic disorder, bipolar disorder, obsessive compulsive disorder, bulimia nervosa, or anorexia nervosa in the 3 months prior to the screening; any substance use disorder (except for nicotine or caffeine use disorder).
* Patients who, in the investigator's judgment, pose a current, serious suicidal or homicidal risk
* Presence of a serious or unstable medical illness, including insulin-dependent diabetes mellitus or bleeding disorder which, in the investigator's opinion, could compromise response to treatment, participant safety, or interpretation of study results.
* Currently breastfeeding, pregnant women, or women of childbearing ability, who do NOT agree to use a study approved method of birth control (described in the MOP) for the duration of the study.
* Currently or within 90 days of screen participating in another clinical trial (excluding large natural cohort trials such as 'All of Us').

Treatment and Concomitant Medication Exclusions:

* Failure to respond during the course of the current major depressive episode to >5 adequate antidepressant trials
* Current use of antipsychotic medications or lithium
* Having received ketamine therapy within 90 days of the screening visit
* Patients who have initiated psychotherapy ≤ 90 days prior to screening.Having received electroconvulsive therapy during the current depressive episode or within 6 months of the screening visit
* Concomitant use of any psychotropic agents within 2 weeks of the baseline visit, except for the ongoing antidepressant, prescription hypnotics, diphenhydramine, or a stable daily dose of a benzodiazepine.
* Concomitant medications that might confound the biomarker findings within 1 week of the baseline visit and during the trial, including: regular (i.e. more than three times per week) ingestion of non-steroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase (COX)-2 inhibitors; any use of oral steroids, immunosuppressants, interferon, chemotherapy, or anticoagulants.

Omega-3 Exclusions:

* A history of severe sensitivity to soy products, fish products, or PUFA supplements
* Patients who had taken supplements enriched with n-3 fatty acids within 60 days of the screening visit or who, at baseline, were consuming a diet containing > 3 g/day of n-3 fatty acids, or who consume > 2 meals of fatty fish per week.
* Having taken a supplement of ≥1 g/day of n-3 fatty acids for ≥6 weeks during the current major depressive episode
* Patients who have had either a poor response or intolerable side effects from n-3s in the past.
* Patients with the following conditions: - Patients with the following conditions: history of atrial fibrillation or atrial flutter, left ventricle hypertrophy, stroke, cardiovascular disease (including coronary artery disease, heart failure, and moderate or severe valve disease or prior valve procedure), uncontrolled hypertension, Crohn's disease, Irritable Bowel Syndrome-diarrhea type, history of gastric bypass surgery, history of cholecystectomy, recent/current history of bulimia with purging, use of prokinetic medications that affect GI transit time, and small intestinal bacterial overgrowth (SIBO)
* Sustained atrial fibrillation or atrial flutter of greater than 30 seconds detected by Holter monitor between V1 (screen) and V2 (baseline)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
18-HEPE (18-hydroxy eicosapentaeoic acid) Change | 12 weeks
  Evaluate change in plasma 18-HEPE (18-hydroxy eicosapentaeoic acid) levels associated with 12 weeks of 4 g/day EPA-enriched n-3 treatment vs placebo.

SECONDARY OUTCOMES:
18-HEPE (18-hydroxy eicosapentaeoic acid) Change in Treatment Responders | 12 weeks
  To evaluate changes in plasma 18-HEPE (18-hydroxy eicosapentaeoic acid) level in relation to sustained clinical response status on the MADRS measure of depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Rapaport, MD, Principal Investigator — University of Utah
Locations (3):
- United States (3):
  - Emory University School of Medicine, Atlanta, Georgia
  - Depression Clinical and Research Program at Massachusetts General Hospital, Boston, Massachusetts
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Data will be stored password-protected in REDCap. Following publication, data will be available to external researchers upon request for replication or secondary analysis. Subject confidentiality will be protected per HIPAA policies. Internal and external requests will be handled by the PI to ensure equitable access, fairness and safeguards. After reviewing a proposal from an external investigator, PI will approve requests with appropriate experimental design, scientific merit and IRB approval and recommend revisions if necessary. Database searches are completed by the study statistician following PI approval, and reports will be provided to investigators. Information can be printed directly from database or exported in spreadsheets in various formats. Format will be controlled by the study statistician. Distribution of data is controlled and de-identified as much as possible.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Following publication of main study findings.
Access Criteria: Interested investigators should contact the study team to inquire about data availability.

REFERENCES:
- [Background] Mischoulon D, Dunlop BW, Kinkead B, Schettler PJ, Lamon-Fava S, Rakofsky JJ, Nierenberg AA, Clain AJ, Mletzko Crowe T, Wong A, Felger JC, Sangermano L, Ziegler TR, Cusin C, Fisher LB, Fava M, Rapaport MH. Omega-3 Fatty Acids for Major Depressive Disorder With High Inflammation: A Randomized Dose-Finding Clinical Trial. J Clin Psychiatry. 2022 Aug 22;83(5):21m14074. doi: 10.4088/JCP.21m14074. PMID 36005883